CLINICAL TRIAL: NCT04999254
Title: Osteopathic Consultation in the Emergency Department for Fresh Lateral Ligament Sprain : a Randomized Controlled Trial
Brief Title: Osteopathic Consultation in the Emergency Department for Fresh Lateral Ligament Sprain
Acronym: OASED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PO21093*
Record Dates: First submitted 2021-08-05; First posted 2021-08-10 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Ankle Sprains
MeSH Terms: conditions — Ankle Injuries | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: participants will be assigned to one of two or more groups in parallel for the duration pot the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic treatment / Usual care (Experimental): osteopathic treatment will be applied in this intervention group.
  Interventions: Other: Medical treatment; Other: osteopathic treatment
- Usual care (Active Comparator): Classic medical treatment
  Interventions: Other: Medical treatment

INTERVENTIONS:
Other: Medical treatment — Medical treatment will be based on functional treatment and the doctor will prescribe the RICE protocol. For this, the patient will have to :
  * place an ice pack on the sprain
  * apply sports rest for three weeks
  * compress the sprain with a compression stocking when standing in order to prevent phlebitis. In addition, to avoid this complication, the doctor will prescribe an anticoagulant.
  * raise the foot with crutches during the day
  * elevate the foot at night or when doing an activity in a sitting position, using a cushion for example.
  In addition, the doctor will prescribe anti-inflammatory drugs to ease the pain and physiotherapy to establish proprioception, muscle strength, joint range and dynamic postural balance of the sprain.
Other: osteopathic treatment — Each patient will be treated as a whole and within a time limit of 45 minutes. The consultation will start with a medical history followed by medical tests. Then, the osteopath will perform osteopathic tests and manual treatment.
  Arms: Osteopathic treatment / Usual care

SUMMARY:
The study consists in recruiting patients with ankle sprains who visit the emergency department (ED).

Each patient will be tested by an osteopath who we will measure pain, swelling and/or edema, and mobility of the ankle. Patients will be asked to reproduce exercises such as to hold on one foot, to stand on tiptoes...

Then, patients will be divided into two groups. The first group will undergo medical treatment during the ED visit, while the second group will undergo osteopathic treatment.

Three time points will be planned. The first one will be the patient's consultation in the ED where treatment will be carried out according to its assignment, as well as the clinical measures previously described. The second time point will be seven days later (plus or minus three days), where only clinical measurements will be performed. The third time point will be three weeks later (plus or minus three days), when the ankle sprain has consolidated, in order to carry out the clinical measurements again.

These clinical measurements will allow to evaluate the effectiveness of a single osteopathic consultation in the ED. The investigators expect a reduction in immediate pain, and thereafter, a reduction in swelling, and an improved mobility and stability of the ankle.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Unilateral sprain
* Stage 1 or 2 sprain
* Recent sprain < 72 hours
* With or without the presence of edema and/or hematoma
* Receiving prior consultation from an ED physician
* Understanding French
* Agreeing to participate in the study and having signed the consent form
* Apyretic
* Patient affiliated to a social security schem

Exclusion Criteria:

* Fractured foot, tibia, fibula
* Stage 3 ankle sprain
* Operated sprain
* Current use of drugs/alcohol
* Altered mental state
* Chronic ankle injury on the contralateral side
* Person deprived of liberty by a judicial or administrative decision
* Neoplasia
* Any contraindication to osteopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-28 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Ankle mobility | Week 3
  measure ankle dorsiflexion range of motion - the injured ankle should have identical mobility to the healthy one

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided